CLINICAL TRIAL: NCT00512135
Title: A Prospective, Open-label, Multicenter, Repeat-dose Trial to Investigate the Safety and Efficacy of NT 201, Free of Complexing Proteins, in the Treatment of Glabellar Frown Lines
Brief Title: Safety and Efficacy of NT 201 (IncobotulinumtoxinA [Xeomin]) in the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 60201-0609/1; 2006-005342-36 (EudraCT Number)
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IncobotulinumtoxinA (Xeomin) (20 units) (Experimental): IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins' (active ingredient: Clostridium Botulinum neurotoxin type A free from complexing proteins) powder for solution for injection; dose: one injection session of solution, prepared by reconstitution of powder with 0.9% sodium chloride (NaCl), 20 units, total volume 0.5 mL, mode of administration: intramuscular injection
  Interventions: Drug: IncobotulinumtoxinA (Xeomin) (20 units)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (Xeomin) (20 units) — Injection of a total of 20 Units incobotulinumtoxinA (Xeomin) on day one of each of up to eight cycles, reconstituted in a total injection volume of 0.5 mL administered in five equal parts of 0.1 mL to five predefined points of the glabellar area.
  Other Names: IncobotulinumtoxinA (Xeomin), also known as 'NT 201' or 'Botulinum toxin type A (150 kD), free from complexing proteins (20 units)

SUMMARY:
The study objective was to investigate the safety and efficacy of incobotulinumtoxinA (Xeomin) during repeat dose treatment of glabellar frown lines. 801 participants with moderate to severe glabellar frown lines at maximum frown who completed participation in one of the studies in this program, i.e. MRZ 60201-0520/1, MRZ 60201-0527/1, MRZ 60201-0724/1, or MRZ 60201-0741/1 were eligible to participate in this repeat-dose study.

DETAILED DESCRIPTION:
This was a prospective, multicenter, open-label, non-control group design Phase 3 clinical study. Approximately 880 participants who were to complete former studies in this program (370 participants from studies MRZ 60201-0520/1 (8) and MRZ 60201-0527/1 (8) as well as approximately 510 participants from studies MRZ 60201-0724/1 (10) and MRZ 60201-0741/1) (11) were expected to enroll in this study in 26 centers in the United States, Canada and Germany. Participants with moderate to severe glabellar frown lines at maximum frown who completed participation in one of these four "feeder" studies in the frown line program were eligible to participate in this repeated dose study. Each participant received a dose of 20 units incobotulinumtoxinA (Xeomin) intramuscular injection on Visit 1 (Day 0 of Cycle 1). Re-injections with 20 U NT 201 could be performed on Day 0 of a subsequent cycle for up to 8 cycles (one cycle >= 85 days). Intervals between treatments were at least three months or 12 weeks, i.e., >= 85 days. For a new treatment cycle to start, the participant had to request a re-injection. The investigator then had to assess if the glabellar frown lines had relapsed to 'moderate' or 'severe'. In this case, a new injection could be administered. The treatment duration per participant was 24 months and up to eight cycles for participants enrolled from studies MRZ 60201-0520/1 and MRZ 60201-0527/1 and 6 months and up to two cycles for participants enrolled from studies MRZ 60201-0724/1 and MRZ 60201-0741/1, respectively. Participants enrolled from studies MRZ 60201-0520/1 and MRZ 60201-0527/1 participated at least one year in the study whereas participants enrolled from studies MRZ 60201-0724/1 and MRZ 60201-0741/1 participated for six months and up to two cycles.

ELIGIBILITY:
Inclusion Criteria:

Participants with 'moderate' or 'severe' glabellar frown lines at maximum frown at the beginning of each treatment cycle (as assessed by the investigator according to FWS) , stable medical condition; Completion of one former study in the Merz NT 201 glabellar program

Exclusion Criteria:

Participants with preexisting neuromuscular diseases (e.g. myasthenia gravis, Lambert-Eaton syndrome) putting the participant at risk, History of Facial Nerve Palsy, Previous treatment with Botulinum Toxin in the glabellar area during the last 12 months, Previous treatment with biodegradable fillers or other procedures (e.g. chemical peeling, photo rejuvenation) in the glabellar area during the last 12 months, Previous insertion of permanent material in the glabellar area; Planned treatment with Botulinum toxin of any serotype in any body region during the study period, Any other planned facial aesthetic procedure in the glabellar area during the trial period; Any surgery in the glabellar area including surgical removal of the corrugator, procerus or depressor supercili muscles or a combination of these or scars in the glabellar area, Inability to substantially lessen glabellar frown lines even by physically spreading apart, Marked facial asymmetry or ptosis of eyelid and/or eyebrow; Any infection in the area of the injection sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2007-06-18 (Actual); Primary Completion 2009-12-28 (Actual); Study Completion 2009-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Rzany, Prof. Dr. med Sc.M., Principal Investigator — Division of Evidence Based Medicine dEBM, Department of Dermatology, Venerology and Allergology , Charité - University Medicine, Berlin, Germany; Timothy Corcoran Flynn, MD, Principal Investigator
Locations (25):
- United States (13):
  - Skin Care Centre, Los Angeles, California
  - About Skin Dermatology, Englewood, Colorado
  - Centre for Cosmetic Enhancement, Aventura, Florida
  - Brandt, Coral Gables, Florida
  - Advanced Dermatology Research Institute, Lincolnshire, Illinois
  - Laser &Skin Surgery Center of Indiana, Carmel, Indiana
  - Coleman, Metairie, Louisiana
  - Skin Care Physisians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Schlessinger, Omaha, Nebraska
  - Image Dermatology P.C., Montclair, New Jersey
  - Narins, White Plains, New York
  - Flynn Consulting PLLC, Raleigh, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
- Canada (2):
  - Carruthers Dermatology Centre Inc., Vancouver, British Columbia
  - Solish, Toronto, Ontario
- Germany (10):
  - Charité Berlin - Klinik für Dermatologie, Berlin
  - Rosenparkklinik, Darmstadt
  - Krankenhaus Dresden Friedrichstadt, Dresden
  - Johann-Wolfgang-Goethe- Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universität Hamburg, Hamburg
  - SCIderm GmbH, Hamburg
  - Uniklinik Saarland, Homburg / Saar
  - Dr. Michael Sebastian, Mahlow
  - Dr. Hans-Ulrich Voigt, München
  - Dr. Thomas Dirschka, Wuppertal

REFERENCES:
- [Result] Rzany B, Flynn TC, Schlobe A, Heinz M, Harrington L. Long-term results for incobotulinumtoxinA in the treatment of glabellar frown lines. Dermatol Surg. 2013 Jan;39(1 Pt 1):95-103. doi: 10.1111/dsu.12008. Epub 2012 Nov 27. PMID 23190342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderate to severe glabellar frown lines at maximum frown who completed one of the four feeder studies MRZ 60201-0520/1 (NCT00430963), MRZ 60201-0527/1 (NCT00430586), MRZ 60201-0724/1 (NCT00512135), or MRZ 60201-0741/1(NCT00512135) were enrolled in this repeat-dose study at 26 investigational sites in the United States, Canada and Germany.
Pre-assignment Details: A total of 810 participants were screened, out of which 801 were enrolled into the study. Of these 801 participants, 796 received the study treatment.
Groups:
- IncobotulinumtoxinA 20 U: Participants, pre-treated with placebo, and incobotulinumtoxinA (NT 201) 10, 20 and 30 units (U) in feeder studies; received incobotulinumtoxinA 20 U powder for solution for injection, intramuscularly, in equal aliquots to 5 injection sites (Point A [one injection in procerus muscle at crossing of two lines that connect Point B and contralateral caruncle], Point B [one injection on each side in central part of corrugator muscle approximately 1 centimeter (cm) above bony orbital rim on an imaginary line drawn vertically from caruncle], and Point C [one injection on each side in middle part of corrugator muscle at least 1.5 cm above bony orbital rim on an imaginary line drawn vertically from midpupillary line]) on Day 0 of Cycle 1. Re-injections based on investigator assessment were performed on Day 0 of subsequent cycles (up to 8 cycles for participants enrolled from MRZ 60201-0520/1 and MRZ 60201-0527/1; and up to 2 cycles for participants enrolled from MRZ 60201-0724/1 and MRZ 60201-0741/1). Each cycle length greater than or equal to (>=) 85 days.
Period: Overall Study
Arm/Group | IncobotulinumtoxinA 20 U
Started | 801
Treated | 796
Completed | 717
Not Completed | 84
Not completed — Not Treated | 5
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 27
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were successfully screened for the study (signed the Informed Consent form [ICF]) and received at least one injection of the study drug.
Groups:
- IncobotulinumtoxinA 20 U: Participants, pre-treated with placebo, and incobotulinumtoxinA (NT 201) 10, 20 and 30 U in feeder studies; received incobotulinumtoxinA 20 U powder for solution for injection, intramuscularly, in equal aliquots to 5 injection sites (Point A [one injection in procerus muscle at crossing of two lines that connect Point B and contralateral caruncle], Point B [one injection on each side in central part of corrugator muscle approximately 1 cm) above bony orbital rim on an imaginary line drawn vertically from caruncle], and Point C [one injection on each side in middle part of corrugator muscle at least 1.5 cm above bony orbital rim on an imaginary line drawn vertically from midpupillary line]) on Day 0 of Cycle 1. Re-injections based on investigator assessment were performed on Day 0 of subsequent cycles (up to 8 cycles for participants enrolled from MRZ 60201-0520/1 and MRZ 60201-0527/1; and up to 2 cycles for participants enrolled from MRZ 60201-0724/1 and MRZ 60201-0741/1). Each cycle length >=85 days.
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702
  Male | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 26
  Black or African American | 10
  Hispanic or Latino | 81
  Native Hawaiian or Other Pacific Islander | 0
  White | 669
  Other | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 177
  North America | 619

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Baseline up to Month 30
Population: The FAS consisted of all participants who were successfully screened for the study (signed the ICF) and received at least one injection of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- IncobotulinumtoxinA 20 U: Participants, pre-treated with placebo, and incobotulinumtoxinA (NT 201) 10, 20 and 30 U in feeder studies; received incobotulinumtoxinA 20 U powder for solution for injection, intramuscularly, in equal aliquots to 5 injection sites (Point A [one injection in procerus muscle at crossing of two lines that connect Point B and contralateral caruncle], Point B [one injection on each side in central part of corrugator muscle approximately 1 cm above bony orbital rim on an imaginary line drawn vertically from caruncle], and Point C [one injection on each side in middle part of corrugator muscle at least 1.5 cm above bony orbital rim on an imaginary line drawn vertically from midpupillary line]) on Day 0 of Cycle 1. Re-injections based on investigator assessment were performed on Day 0 of subsequent cycles (up to 8 cycles for participants enrolled from MRZ 60201-0520/1 and MRZ 60201-0527/1; and up to 2 cycles for participants enrolled from MRZ 60201-0724/1 and MRZ 60201-0741/1). Each cycle length >=85 days.
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
Participants | 374

2. Primary Outcome: Incidence of Adverse Events of Special Interest (AESI)
Time Frame: Baseline up to Month 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
Participants | 9

3. Primary Outcome: Percentage of Responders at Maximum Frown as Assessed by the Investigator According to Facial Wrinkle Scale (FWS)
Description: FWS was used to assess the severity of glabellar frown lines at maximum frown by the investigator. The 4-point scale depicted as: 0 = none, 1 = mild, 2 = moderate and 3 = severe. Responders on the FWS were defined as participants with glabellar line severity of none (0) or mild (1).
Time Frame: At evaluation visit (30 days after injection) and at last control visit (85 days after last injection) in each treatment cycle from Cycle 1 to Cycle 8 (each cycle length >=85 days)
Population: The FAS consisted of all participants who were successfully screened for the study (signed the ICF) and received at least one injection of the study drug. Here number analyzed "n" were the participants who were evaluable for this outcome measure at given time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
percentage of participants
  Cycle 1: Evaluation Visit | 79.1 [76.2 to 81.8]
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 694
  Cycle 2: Evaluation Visit | 79.8 [76.7 to 82.6]
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 322
  Cycle 3: Evaluation Visit | 80.1 [75.4 to 84.1]
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 309
  Cycle 4: Evaluation Visit | 80.3 [75.5 to 84.3]
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 291
  Cycle 5: Evaluation Visit | 81.4 [76.6 to 85.5]
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 261
  Cycle 6: Evaluation Visit | 81.2 [76.0 to 85.5]
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 191
  Cycle 7: Evaluation Visit | 82.7 [76.7 to 87.4]
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit | 89.6 [77.8 to 95.5]
  Cycle 1: Last Control Visit | 6.5 [5.0 to 8.5]
  Cycle 2: Last Control Visit: number analyzed (Participants) | 694
  Cycle 2: Last Control Visit | 16.6 [14.0 to 19.5]
  Cycle 3: Last Control Visit: number analyzed (Participants) | 322
  Cycle 3: Last Control Visit | 0.6 [0.2 to 2.2]
  Cycle 4: Last Control Visit: number analyzed (Participants) | 309
  Cycle 4: Last Control Visit | 0.6 [0.2 to 2.3]
  Cycle 5: Last Control Visit: number analyzed (Participants) | 291
  Cycle 5: Last Control Visit | 4.8 [2.9 to 7.9]
  Cycle 6: Last Control Visit: number analyzed (Participants) | 261
  Cycle 6: Last Control Visit | 8.8 [5.9 to 12.9]
  Cycle 7: Last Control Visit: number analyzed (Participants) | 191
  Cycle 7: Last Control Visit | 17.8 [13.0 to 23.8]
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit | 29.2 [18.2 to 43.2]

4. Primary Outcome: Percentage of Responders at Rest as Assessed by the Investigator According to FWS
Description: FWS was used to assess the severity of glabellar frown lines at rest by the investigator. The 4-point scale depicted as: 0 = none, 1 = mild, 2 = moderate and 3 = severe. Responders on the FWS were defined as participants with glabellar line severity of none (0) or mild (1). Responders on the FWS were defined as participants with glabellar line severity of none (0) or mild (1).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
percentage of participants
  Cycle 1: Evaluation Visit | 78.9 [75.9 to 81.6]
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 694
  Cycle 2: Evaluation Visit | 79.7 [76.5 to 82.5]
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 322
  Cycle 3: Evaluation Visit | 80.7 [76.1 to 84.7]
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 309
  Cycle 4: Evaluation Visit | 80.6 [75.8 to 84.6]
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 291
  Cycle 5: Evaluation Visit | 79.4 [74.4 to 83.6]
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 261
  Cycle 6: Evaluation Visit | 77.0 [71.5 to 81.7]
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 191
  Cycle 7: Evaluation Visit | 81.2 [75.0 to 86.1]
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit | 87.5 [75.3 to 94.1]
  Cycle 1: Last Control Visit | 57.0 [53.6 to 60.4]
  Cycle 2: Last Control Visit: number analyzed (Participants) | 694
  Cycle 2: Last Control Visit | 63.8 [60.2 to 67.3]
  Cycle 3: Last Control Visit: number analyzed (Participants) | 322
  Cycle 3: Last Control Visit | 63.7 [58.3 to 68.7]
  Cycle 4: Last Control Visit: number analyzed (Participants) | 309
  Cycle 4: Last Control Visit | 60.5 [55.0 to 65.8]
  Cycle 5: Last Control Visit: number analyzed (Participants) | 291
  Cycle 5: Last Control Visit | 63.2 [57.6 to 68.6]
  Cycle 6: Last Control Visit: number analyzed (Participants) | 261
  Cycle 6: Last Control Visit | 64.4 [58.4 to 69.9]
  Cycle 7: Last Control Visit: number analyzed (Participants) | 191
  Cycle 7: Last Control Visit | 67.0 [60.1 to 73.3]
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit | 83.3 [70.4 to 91.3]

5. Primary Outcome: Percentage of Responders at Maximum Frown by Participant's Assessment on the 4-point Scale
Description: Participant's assessment of the glabellar frown lines at maximum frown on the 4-point scale was done by asking participant the following question in local language: "How would you judge the potency of frown muscle action by comparison to sample photos at this visit?" The possible rating responses were: 0 = no muscle action at all, 1 = some even slight muscle action possible, 2 = moderately strong muscle action possible, 3 = strong muscle action possible which may cause local pallor. Responders were participants with at least 1-point improvement compared to Day 0 whereas improvement was expressed by lowering of the numerical score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
percentage of participants
  Cycle 1: Evaluation Visit | 86.2 [83.6 to 88.4]
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 694
  Cycle 2: Evaluation Visit | 87.6 [84.9 to 89.9]
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 322
  Cycle 3: Evaluation Visit | 88.2 [84.2 to 91.3]
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 309
  Cycle 4: Evaluation Visit | 87.4 [83.2 to 90.6]
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 291
  Cycle 5: Evaluation Visit | 85.9 [81.4 to 89.4]
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 261
  Cycle 6: Evaluation Visit | 88.5 [84.1 to 91.8]
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 191
  Cycle 7: Evaluation Visit | 90.1 [85.0 to 93.5]
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit | 93.8 [83.2 to 97.9]
  Cycle 1: Last Control Visit | 31.2 [28.0 to 34.5]
  Cycle 2: Last Control Visit: number analyzed (Participants) | 694
  Cycle 2: Last Control Visit | 43.8 [40.2 to 47.5]
  Cycle 3: Last Control Visit: number analyzed (Participants) | 322
  Cycle 3: Last Control Visit | 38.2 [33.1 to 43.6]
  Cycle 4: Last Control Visit: number analyzed (Participants) | 309
  Cycle 4: Last Control Visit | 37.9 [32.6 to 43.4]
  Cycle 5: Last Control Visit: number analyzed (Participants) | 291
  Cycle 5: Last Control Visit | 43.6 [38.1 to 49.4]
  Cycle 6: Last Control Visit: number analyzed (Participants) | 261
  Cycle 6: Last Control Visit | 41.8 [35.9 to 47.8]
  Cycle 7: Last Control Visit: number analyzed (Participants) | 191
  Cycle 7: Last Control Visit | 52.4 [45.3 to 59.3]
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit | 60.4 [46.3 to 73.0]

6. Primary Outcome: Percentage of Responders at Rest by Participant's Assessment on the 4-point Scale
Description: Participant's assessment of the glabellar frown lines at rest on the 4-point scale was done by asking participant the following question in local language: "How would you judge the degree of your glabellar lines by comparison to sample photos at this visit?" The possible rating responses were: 0 = no visible vertical line(s) at all, 1 = slightly visible vertical line(s), 2 = moderate vertical line(s) with depression, and 3 = deep vertical line(s) and depression which cannot be effaced by spreading. Responders were participants with at least 1-point improvement compared to Day 0 whereas improvement was expressed by lowering of the numerical score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 796
percentage of participants
  Cycle 1: Evaluation Visit | 69.5 [66.2 to 72.6]
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 694
  Cycle 2: Evaluation Visit | 67.0 [63.4 to 70.4]
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 322
  Cycle 3: Evaluation Visit | 73.0 [67.9 to 77.5]
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 309
  Cycle 4: Evaluation Visit | 73.8 [68.6 to 78.4]
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 291
  Cycle 5: Evaluation Visit | 77.0 [71.8 to 81.4]
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 261
  Cycle 6: Evaluation Visit | 75.1 [69.5 to 80.0]
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 191
  Cycle 7: Evaluation Visit | 75.9 [69.4 to 81.4]
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit | 77.1 [63.5 to 86.7]
  Cycle 1: Last Control Visit | 35.1 [31.8 to 38.4]
  Cycle 2: Last Control Visit: number analyzed (Participants) | 694
  Cycle 2: Last Control Visit | 43.2 [39.6 to 46.9]
  Cycle 3: Last Control Visit: number analyzed (Participants) | 322
  Cycle 3: Last Control Visit | 38.8 [33.7 to 44.2]
  Cycle 4: Last Control Visit: number analyzed (Participants) | 309
  Cycle 4: Last Control Visit | 42.1 [36.7 to 47.6]
  Cycle 5: Last Control Visit: number analyzed (Participants) | 291
  Cycle 5: Last Control Visit | 43.6 [38.1 to 49.4]
  Cycle 6: Last Control Visit: number analyzed (Participants) | 261
  Cycle 6: Last Control Visit | 49.0 [43.0 to 55.1]
  Cycle 7: Last Control Visit: number analyzed (Participants) | 191
  Cycle 7: Last Control Visit | 54.5 [47.4 to 61.4]
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit | 58.3 [44.3 to 71.2]

7. Primary Outcome: Degree of Glabellar Lines as Assessed by the Participant on the 6-point Likert Type Scale at Maximum Frown
Description: Number of participants are reported categorized in grades based on the assessment of the glabellar frown lines at maximum frown on the 6-point Likert scale. Participant's assessment of the glabellar frown lines at maximum frown on the 6-point Likert type scale was done by asking participant the following question in local language: "How would you judge the potency of frown muscle action at this visit?" The possible rating responses were given on a categorical scale of 6 grades between the grades 0 = none at all and 5 = very deep, with higher score reflecting higher potency.
Time Frame: At evaluation visit (30 days after injection); and at last control visit (85 days after last injection) in each treatment cycle from Cycle 1 to Cycle 8 (each cycle length >=85 days)
Population: The FAS consisted of all participants who were successfully screened for the study (signed the ICF) and received at least one injection of the study drug. Here "overall participants analyzed" are participants who were available for this outcome measure assessment and number analyzed "n" were the participants who were evaluable for this outcome measure at given time categories.
Measure: Count of Participants; unit: Participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 786
Participants
  Cycle 1: Evaluation Visit: Grade 0 | 118
  Cycle 1: Evaluation Visit: Grade 1 | 256
  Cycle 1: Evaluation Visit: Grade 2 | 210
  Cycle 1: Evaluation Visit: Grade 3 | 140
  Cycle 1: Evaluation Visit: Grade 4 | 46
  Cycle 1: Evaluation Visit: Grade 5 | 16
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 690
  Cycle 2: Evaluation Visit: Grade 0 | 99
  Cycle 2: Evaluation Visit: Grade 1 | 228
  Cycle 2: Evaluation Visit: Grade 2 | 187
  Cycle 2: Evaluation Visit: Grade 3 | 114
  Cycle 2: Evaluation Visit: Grade 4 | 39
  Cycle 2: Evaluation Visit: Grade 5 | 23
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 319
  Cycle 3: Evaluation Visit: Grade 0 | 52
  Cycle 3: Evaluation Visit: Grade 1 | 113
  Cycle 3: Evaluation Visit: Grade 2 | 84
  Cycle 3: Evaluation Visit: Grade 3 | 44
  Cycle 3: Evaluation Visit: Grade 4 | 19
  Cycle 3: Evaluation Visit: Grade 5 | 7
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 305
  Cycle 4: Evaluation Visit: Grade 0 | 57
  Cycle 4: Evaluation Visit: Grade 1 | 96
  Cycle 4: Evaluation Visit: Grade 2 | 83
  Cycle 4: Evaluation Visit: Grade 3 | 49
  Cycle 4: Evaluation Visit: Grade 4 | 16
  Cycle 4: Evaluation Visit: Grade 5 | 4
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 290
  Cycle 5: Evaluation Visit: Grade 0 | 51
  Cycle 5: Evaluation Visit: Grade 1 | 98
  Cycle 5: Evaluation Visit: Grade 2 | 84
  Cycle 5: Evaluation Visit: Grade 3 | 35
  Cycle 5: Evaluation Visit: Grade 4 | 19
  Cycle 5: Evaluation Visit: Grade 5 | 3
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 259
  Cycle 6: Evaluation Visit: Grade 0 | 44
  Cycle 6: Evaluation Visit: Grade 1 | 95
  Cycle 6: Evaluation Visit: Grade 2 | 64
  Cycle 6: Evaluation Visit: Grade 3 | 39
  Cycle 6: Evaluation Visit: Grade 4 | 14
  Cycle 6: Evaluation Visit: Grade 5 | 3
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 190
  Cycle 7: Evaluation Visit: Grade 0 | 25
  Cycle 7: Evaluation Visit: Grade 1 | 74
  Cycle 7: Evaluation Visit: Grade 2 | 49
  Cycle 7: Evaluation Visit: Grade 3 | 32
  Cycle 7: Evaluation Visit: Grade 4 | 9
  Cycle 7: Evaluation Visit: Grade 5 | 1
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit: Grade 0 | 5
  Cycle 8: Evaluation Visit: Grade 1 | 22
  Cycle 8: Evaluation Visit: Grade 2 | 14
  Cycle 8: Evaluation Visit: Grade 3 | 5
  Cycle 8: Evaluation Visit: Grade 4 | 1
  Cycle 8: Evaluation Visit: Grade 5 | 1
  Cycle 1: Last Control Visit: number analyzed (Participants) | 777
  Cycle 1: Last Control Visit: Grade 0 | 6
  Cycle 1: Last Control Visit: Grade 1 | 28
  Cycle 1: Last Control Visit: Grade 2 | 99
  Cycle 1: Last Control Visit: Grade 3 | 223
  Cycle 1: Last Control Visit: Grade 4 | 259
  Cycle 1: Last Control Visit: Grade 5 | 162
  Cycle 2: Last Control Visit: number analyzed (Participants) | 681
  Cycle 2: Last Control Visit: Grade 0 | 9
  Cycle 2: Last Control Visit: Grade 1 | 54
  Cycle 2: Last Control Visit: Grade 2 | 97
  Cycle 2: Last Control Visit: Grade 3 | 208
  Cycle 2: Last Control Visit: Grade 4 | 208
  Cycle 2: Last Control Visit: Grade 5 | 105
  Cycle 3: Last Control Visit: number analyzed (Participants) | 317
  Cycle 3: Last Control Visit: Grade 0 | 0
  Cycle 3: Last Control Visit: Grade 1 | 10
  Cycle 3: Last Control Visit: Grade 2 | 49
  Cycle 3: Last Control Visit: Grade 3 | 100
  Cycle 3: Last Control Visit: Grade 4 | 114
  Cycle 3: Last Control Visit: Grade 5 | 44
  Cycle 4: Last Control Visit: number analyzed (Participants) | 304
  Cycle 4: Last Control Visit: Grade 0 | 0
  Cycle 4: Last Control Visit: Grade 1 | 14
  Cycle 4: Last Control Visit: Grade 2 | 41
  Cycle 4: Last Control Visit: Grade 3 | 104
  Cycle 4: Last Control Visit: Grade 4 | 90
  Cycle 4: Last Control Visit: Grade 5 | 55
  Cycle 5: Last Control Visit: number analyzed (Participants) | 287
  Cycle 5: Last Control Visit: Grade 0 | 1
  Cycle 5: Last Control Visit: Grade 1 | 16
  Cycle 5: Last Control Visit: Grade 2 | 55
  Cycle 5: Last Control Visit: Grade 3 | 89
  Cycle 5: Last Control Visit: Grade 4 | 81
  Cycle 5: Last Control Visit: Grade 5 | 45
  Cycle 6: Last Control Visit: number analyzed (Participants) | 257
  Cycle 6: Last Control Visit: Grade 0 | 2
  Cycle 6: Last Control Visit: Grade 1 | 16
  Cycle 6: Last Control Visit: Grade 2 | 52
  Cycle 6: Last Control Visit: Grade 3 | 73
  Cycle 6: Last Control Visit: Grade 4 | 83
  Cycle 6: Last Control Visit: Grade 5 | 31
  Cycle 7: Last Control Visit: number analyzed (Participants) | 189
  Cycle 7: Last Control Visit: Grade 0 | 3
  Cycle 7: Last Control Visit: Grade 1 | 16
  Cycle 7: Last Control Visit: Grade 2 | 50
  Cycle 7: Last Control Visit: Grade 3 | 51
  Cycle 7: Last Control Visit: Grade 4 | 52
  Cycle 7: Last Control Visit: Grade 5 | 17
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit: Grade 0 | 0
  Cycle 8: Last Control Visit: Grade 1 | 4
  Cycle 8: Last Control Visit: Grade 2 | 14
  Cycle 8: Last Control Visit: Grade 3 | 13
  Cycle 8: Last Control Visit: Grade 4 | 13
  Cycle 8: Last Control Visit: Grade 5 | 4

8. Primary Outcome: Degree of Glabellar Lines as Assessed by the Participant on the 6-point Likert Type Scale at Rest
Description: Number of participants are reported categorized in grades based on the assessment of the glabellar frown lines at rest on the 6-point Likert scale. Participant's assessment of the glabellar frown lines at rest on the 6-point Likert type scale was done by asking participant the following question in local language: "How would you judge the degree of your glabellar lines at this visit?" The possible rating responses were given on a categorical scale of 6 grades between the grades 0 = none at all and 5 = very deep, with higher scores reflecting higher degree of glabellar lines.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 786
Participants
  Cycle 1: Evaluation Visit: Grade 0 | 237
  Cycle 1: Evaluation Visit: Grade 1 | 281
  Cycle 1: Evaluation Visit: Grade 2 | 144
  Cycle 1: Evaluation Visit: Grade 3 | 89
  Cycle 1: Evaluation Visit: Grade 4 | 28
  Cycle 1: Evaluation Visit: Grade 5 | 7
  Cycle 2: Evaluation Visit: number analyzed (Participants) | 690
  Cycle 2: Evaluation Visit: Grade 0 | 205
  Cycle 2: Evaluation Visit: Grade 1 | 251
  Cycle 2: Evaluation Visit: Grade 2 | 150
  Cycle 2: Evaluation Visit: Grade 3 | 57
  Cycle 2: Evaluation Visit: Grade 4 | 15
  Cycle 2: Evaluation Visit: Grade 5 | 12
  Cycle 3: Evaluation Visit: number analyzed (Participants) | 319
  Cycle 3: Evaluation Visit: Grade 0 | 98
  Cycle 3: Evaluation Visit: Grade 1 | 111
  Cycle 3: Evaluation Visit: Grade 2 | 72
  Cycle 3: Evaluation Visit: Grade 3 | 29
  Cycle 3: Evaluation Visit: Grade 4 | 5
  Cycle 3: Evaluation Visit: Grade 5 | 4
  Cycle 4: Evaluation Visit: number analyzed (Participants) | 305
  Cycle 4: Evaluation Visit: Grade 0 | 90
  Cycle 4: Evaluation Visit: Grade 1 | 123
  Cycle 4: Evaluation Visit: Grade 2 | 53
  Cycle 4: Evaluation Visit: Grade 3 | 34
  Cycle 4: Evaluation Visit: Grade 4 | 2
  Cycle 4: Evaluation Visit: Grade 5 | 3
  Cycle 5: Evaluation Visit: number analyzed (Participants) | 290
  Cycle 5: Evaluation Visit: Grade 0 | 92
  Cycle 5: Evaluation Visit: Grade 1 | 111
  Cycle 5: Evaluation Visit: Grade 2 | 52
  Cycle 5: Evaluation Visit: Grade 3 | 25
  Cycle 5: Evaluation Visit: Grade 4 | 7
  Cycle 5: Evaluation Visit: Grade 5 | 3
  Cycle 6: Evaluation Visit: number analyzed (Participants) | 259
  Cycle 6: Evaluation Visit: Grade 0 | 80
  Cycle 6: Evaluation Visit: Grade 1 | 102
  Cycle 6: Evaluation Visit: Grade 2 | 55
  Cycle 6: Evaluation Visit: Grade 3 | 13
  Cycle 6: Evaluation Visit: Grade 4 | 6
  Cycle 6: Evaluation Visit: Grade 5 | 3
  Cycle 7: Evaluation Visit: number analyzed (Participants) | 190
  Cycle 7: Evaluation Visit: Grade 0 | 59
  Cycle 7: Evaluation Visit: Grade 1 | 76
  Cycle 7: Evaluation Visit: Grade 2 | 37
  Cycle 7: Evaluation Visit: Grade 3 | 12
  Cycle 7: Evaluation Visit: Grade 4 | 3
  Cycle 7: Evaluation Visit: Grade 5 | 3
  Cycle 8: Evaluation Visit: number analyzed (Participants) | 48
  Cycle 8: Evaluation Visit: Grade 0 | 12
  Cycle 8: Evaluation Visit: Grade 1 | 27
  Cycle 8: Evaluation Visit: Grade 2 | 6
  Cycle 8: Evaluation Visit: Grade 3 | 2
  Cycle 8: Evaluation Visit: Grade 4 | 1
  Cycle 8: Evaluation Visit: Grade 5 | 0
  Cycle 1: Last Control Visit: number analyzed (Participants) | 777
  Cycle 1: Last Control Visit: Grade 0 | 70
  Cycle 1: Last Control Visit: Grade 1 | 204
  Cycle 1: Last Control Visit: Grade 2 | 241
  Cycle 1: Last Control Visit: Grade 3 | 163
  Cycle 1: Last Control Visit: Grade 4 | 71
  Cycle 1: Last Control Visit: Grade 5 | 28
  Cycle 2: Last Control Visit: number analyzed (Participants) | 681
  Cycle 2: Last Control Visit: Grade 0 | 98
  Cycle 2: Last Control Visit: Grade 1 | 199
  Cycle 2: Last Control Visit: Grade 2 | 190
  Cycle 2: Last Control Visit: Grade 3 | 125
  Cycle 2: Last Control Visit: Grade 4 | 50
  Cycle 2: Last Control Visit: Grade 5 | 19
  Cycle 3: Last Control Visit: number analyzed (Participants) | 317
  Cycle 3: Last Control Visit: Grade 0 | 31
  Cycle 3: Last Control Visit: Grade 1 | 81
  Cycle 3: Last Control Visit: Grade 2 | 88
  Cycle 3: Last Control Visit: Grade 3 | 81
  Cycle 3: Last Control Visit: Grade 4 | 24
  Cycle 3: Last Control Visit: Grade 5 | 12
  Cycle 4: Last Control Visit: number analyzed (Participants) | 304
  Cycle 4: Last Control Visit: Grade 0 | 32
  Cycle 4: Last Control Visit: Grade 1 | 88
  Cycle 4: Last Control Visit: Grade 2 | 82
  Cycle 4: Last Control Visit: Grade 3 | 65
  Cycle 4: Last Control Visit: Grade 4 | 30
  Cycle 4: Last Control Visit: Grade 5 | 7
  Cycle 5: Last Control Visit: number analyzed (Participants) | 287
  Cycle 5: Last Control Visit: Grade 0 | 33
  Cycle 5: Last Control Visit: Grade 1 | 71
  Cycle 5: Last Control Visit: Grade 2 | 96
  Cycle 5: Last Control Visit: Grade 3 | 55
  Cycle 5: Last Control Visit: Grade 4 | 25
  Cycle 5: Last Control Visit: Grade 5 | 7
  Cycle 6: Last Control Visit: number analyzed (Participants) | 257
  Cycle 6: Last Control Visit: Grade 0 | 34
  Cycle 6: Last Control Visit: Grade 1 | 73
  Cycle 6: Last Control Visit: Grade 2 | 90
  Cycle 6: Last Control Visit: Grade 3 | 35
  Cycle 6: Last Control Visit: Grade 4 | 20
  Cycle 6: Last Control Visit: Grade 5 | 5
  Cycle 7: Last Control Visit: number analyzed (Participants) | 189
  Cycle 7: Last Control Visit: Grade 0 | 33
  Cycle 7: Last Control Visit: Grade 1 | 64
  Cycle 7: Last Control Visit: Grade 2 | 54
  Cycle 7: Last Control Visit: Grade 3 | 24
  Cycle 7: Last Control Visit: Grade 4 | 10
  Cycle 7: Last Control Visit: Grade 5 | 4
  Cycle 8: Last Control Visit: number analyzed (Participants) | 48
  Cycle 8: Last Control Visit: Grade 0 | 3
  Cycle 8: Last Control Visit: Grade 1 | 24
  Cycle 8: Last Control Visit: Grade 2 | 10
  Cycle 8: Last Control Visit: Grade 3 | 5
  Cycle 8: Last Control Visit: Grade 4 | 6
  Cycle 8: Last Control Visit: Grade 5 | 0

9. Primary Outcome: Time to Onset of Treatment Effect
Description: Onset of treatment effect was analyzed using number of participants with corresponding onset of treatment effect, stratified by cycles.
Time Frame: From injection visit up to date of onset of treatment effect in each treatment cycle from Cycle 1 to Cycle 8 (each cycle length >=85 days)
Population: The FAS consists of all participants who were successfully screened for the study (signed the ICF) and received at least one injection of the study drug. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure and number analyzed "n" were the participants who were evaluable for this outcome measure at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | IncobotulinumtoxinA 20 U
Number analyzed (Participants) | 786
Participants
  Cycle 1: None | 15
  Cycle 1: Day 0 | 10
  Cycle 1: Day 1 | 86
  Cycle 1: Day 2 | 168
  Cycle 1: Day 3 | 171
  Cycle 1: Day 4 | 93
  Cycle 1: Day 5 | 75
  Cycle 1: Day 6 | 33
  Cycle 1: Day 7 | 70
  Cycle 1: Day 8 | 12
  Cycle 1: Day 9 | 5
  Cycle 1: Day >=10 | 48
  Cycle 2: number analyzed (Participants) | 690
  Cycle 2: None | 20
  Cycle 2: Day 0 | 22
  Cycle 2: Day 1 | 106
  Cycle 2: Day 2 | 134
  Cycle 2: Day 3 | 138
  Cycle 2: Day 4 | 82
  Cycle 2: Day 5 | 53
  Cycle 2: Day 6 | 17
  Cycle 2: Day 7 | 58
  Cycle 2: Day 8 | 10
  Cycle 2: Day 9 | 9
  Cycle 2: Day >=10 | 41
  Cycle 3: number analyzed (Participants) | 319
  Cycle 3: None | 6
  Cycle 3: Day 0 | 8
  Cycle 3: Day 1 | 44
  Cycle 3: Day 2 | 56
  Cycle 3: Day 3 | 70
  Cycle 3: Day 4 | 46
  Cycle 3: Day 5 | 36
  Cycle 3: Day 6 | 11
  Cycle 3: Day 7 | 18
  Cycle 3: Day 8 | 3
  Cycle 3: Day 9 | 6
  Cycle 3: Day >=10 | 15
  Cycle 4: number analyzed (Participants) | 305
  Cycle 4: None | 4
  Cycle 4: Day 0 | 10
  Cycle 4: Day 1 | 39
  Cycle 4: Day 2 | 54
  Cycle 4: Day 3 | 78
  Cycle 4: Day 4 | 33
  Cycle 4: Day 5 | 29
  Cycle 4: Day 6 | 6
  Cycle 4: Day 7 | 22
  Cycle 4: Day 8 | 6
  Cycle 4: Day 9 | 6
  Cycle 4: Day >=10 | 18
  Cycle 5: number analyzed (Participants) | 290
  Cycle 5: None | 6
  Cycle 5: Day 0 | 9
  Cycle 5: Day 1 | 37
  Cycle 5: Day 2 | 64
  Cycle 5: Day 3 | 57
  Cycle 5: Day 4 | 39
  Cycle 5: Day 5 | 21
  Cycle 5: Day 6 | 17
  Cycle 5: Day 7 | 20
  Cycle 5: Day 8 | 5
  Cycle 5: Day 9 | 4
  Cycle 5: Day >=10 | 11
  Cycle 6: number analyzed (Participants) | 259
  Cycle 6: None | 2
  Cycle 6: Day 0 | 10
  Cycle 6: Day 1 | 33
  Cycle 6: Day 2 | 46
  Cycle 6: Day 3 | 56
  Cycle 6: Day 4 | 42
  Cycle 6: Day 5 | 20
  Cycle 6: Day 6 | 5
  Cycle 6: Day 7 | 21
  Cycle 6: Day 8 | 7
  Cycle 6: Day 9 | 2
  Cycle 6: Day >=10 | 15
  Cycle 7: number analyzed (Participants) | 190
  Cycle 7: None | 3
  Cycle 7: Day 0 | 8
  Cycle 7: Day 1 | 17
  Cycle 7: Day 2 | 36
  Cycle 7: Day 3 | 43
  Cycle 7: Day 4 | 29
  Cycle 7: Day 5 | 19
  Cycle 7: Day 6 | 8
  Cycle 7: Day 7 | 15
  Cycle 7: Day 8 | 6
  Cycle 7: Day 9 | 1
  Cycle 7: Day >=10 | 5
  Cycle 8: number analyzed (Participants) | 48
  Cycle 8: None | 0
  Cycle 8: Day 0 | 1
  Cycle 8: Day 1 | 6
  Cycle 8: Day 2 | 4
  Cycle 8: Day 3 | 17
  Cycle 8: Day 4 | 4
  Cycle 8: Day 5 | 7
  Cycle 8: Day 6 | 2
  Cycle 8: Day 7 | 4
  Cycle 8: Day 8 | 2
  Cycle 8: Day 9 | 0
  Cycle 8: Day >=10 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Month 30
Description: The investigator asked the participant for AEs systematically at each visit.
Groups:
- IncobotulinumtoxinA 20 U: Participants, pre-treated with placebo, and incobotulinumtoxinA (NT 201) 10, 20 and 30 U in feeder studies; received incobotulinumtoxinA 20 U powder for solution for injection, intramuscularly, in equal aliquots to 5 injection sites (Point A [one injection in procerus muscle at crossing of two lines that connect Point B and contralateral caruncle], Point B [one injection on each side in central part of corrugator muscle approximately 1 cm above bony orbital rim on an imaginary line drawn vertically from caruncle], and Point C [one injection on each side in middle part of corrugator muscle at least 1.5 cm above bony orbital rim on an imaginary line drawn vertically from midpupillary line]) on Day 0 of Cycle 1. Re-injections based on investigator assessment were performed on Day 0 of subsequent cycles (up to 8 cycles for participants enrolled from MRZ 60201-0520/1 and MRZ 60201-0527/1; and up to 2 cycles for participants enrolled from MRZ 60201-0724/1 and MRZ 60201-0741/1). Each cycle length = 90 days.
Arm/Group | IncobotulinumtoxinA 20 U
All-Cause Mortality (participants affected / at risk) | 0/796
Serious Adverse Events (participants affected / at risk) | 29/796
Other Adverse Events (participants affected / at risk) | 169/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA 20 U (N=796)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 2 (2)
Mammoplasty (Surgical and medical procedures) | 2 (2)
Cardiac operation (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Cystopexy (Surgical and medical procedures) | 1 (1)
Phlebectomy (Surgical and medical procedures) | 1 (1)
Polypectomy (Surgical and medical procedures) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (2)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA 20 U (N=796)
Nasopharyngitis (Infections and infestations) | 109 (154)
Headache (Nervous system disorders) | 60 (116)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.